CLINICAL TRIAL: NCT02127203
Title: Assessment of Nitro - Oxidative Stress in Periodontal Disease
Brief Title: Nitro-oxidative Stress in Periodontitis
Status: Completed | Type: Observational
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Other Study IDs: UDDS-Perio-03-2014
Record Dates: First submitted 2014-04-25; First posted 2014-04-30 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Periodontitis; Aggressive Periodontitis
Keywords: oxidative stress; periodontal disease; nitric oxide
MeSH Terms: conditions — Chronic Periodontitis; Aggressive Periodontitis; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Chronic Periodontitis group (ChP): 20 patients aged > 45 years and have presence of ≥2 non-adjacent sites per quadrant that were not first molars or incisors, with probing depth (PD) ≥5 mm, which bleed on gentle probing. The demonstrated radiographic bone loss ≥30% of the root length, patient with poor oral hygiene, the amount of accumulated plaque commensurate with the amount of clinical attachment level (CAL)
- Resistant Control group (R): 20 age-sex matched patients who are > 45 years exhibit no signs of periodontal disease as determined by the absence of the evidence of interproximal (CAL ≤ 1mm), PD > 3 mm at any site, whole-mouth bleeding scores <10% and have no clinical signs of gingival inflammation .
- Aggressive Periodontitis group (AgP): 20 patients who are aged < 35 years and diagnosed with rapid attachment loss with periodontal pocket depth (PD) > 4 mm around at least three teeth other than the first molars and incisors. Rapid bone destruction (>50%bone loss at diseased sites). Weak relationship between dental plaque and the severity of gingival inflammation.
- Young Control group (YC): 20 age- and sex matched patients who are < 35 years and exhibit no signs of periodontal disease.

SUMMARY:
Periodontitis is a chronic inflammatory disease whose etio-pathogencity is not fully understood yet. Reactive oxygen species (ROS) and reactive nitrogen species (RNS) are involved in physiological and pathological processes. Nitro-oxidative stress has been implicated in Periodontitis.

The aim of this study is to assess the levels of ROS and RNS in serum and gingival crevicular fluid (GCF) samples taken from periodontitis (chronic and aggressive) patients and healthy controls. Subsequently, correlating these levels with the severity of periodontal disease.

Eighty subjects will be invited to participate in this study. Patients will be allocated into four groups (20 patients each). The biochemical parameters that will be investigated are Malondialdehyde (MDA) (using TBRSA assay) as a marker of oxidative stress and (NO- level using Griess reagent) as a marker of nitrosative stress.

DETAILED DESCRIPTION:
Introduction:

Teeth and their supporting periodontal structures are of great importance in good oral health. Periodontitis is an inflammatory disease of the periodontium which affects the supporting tissues of the teeth. The disease is multifaceted and its etio-pathogenecity is still not fully understood and therefore the treatment of different types of periodontal disease can be very difficult. Numerous risk factors have been implicated in the disease process including risk determinants and risk indicators. Most recently, strong body of evidence has accumulated to support a role for reactive oxygen (ROS) and nitrogen species (RNS) either as trigger agents or more frequently, aggravators of the primary lesions in periodontitis.

Oxygen and nitrogen reactive species are involved in a large number of physiological and pathological processes. ROS generated by monocytes and neutrophyles during inflammation are important aggression factors in the periodontal tissues. ROS play an important role in activation of osteoclasts and in bone resorption.

Oxidative stress is a condition arising when there is a serious imbalance between the levels of free radicals in a cell and its antioxidant defenses in favor of the former. Thus, tissue damage can result when antioxidant systems are unable to counteract the free radicals actions efficiently. Inflammation when stimulated by bacterial pathogens, host cells release proinflammatory cytokines (IL-1α, IL-6, IL-8, and tumor necrosis factor-α) as part of immune response. These cytokines recruit polymorphonuclear cells (PMNs) that play a major role in the etiology of periodontal disease by producing proteolytic enzymes, such as elastase and O2 (molecular oxygen) by the oxidative burst.

In a recent study, Abou Sulaiman & Shehadeh found that serum total antioxidant capacity (TAS) was lower in non-smokers Syrian patients with chronic periodontitis compared to healthy controls. Also, they reported that periodontal treatment restored TAS levels to normal levels similar to healthy controls.

The aim of this study is to assess the levels of ROS and RNS in serum and gingival crevicular fluid (GCF) samples taken from periodontitis patients (chronic and aggressive) and healthy controls. Subsequently, correlating these levels with severity of periodontal disease in Syrian patients.

Materials and methods:

A total of 80 subjects will be invited to participate in this study from the patients referred to the Department of Periodontology, Faculty of Dentistry, University of Damascus. The study has been approved by our local Review Board. Subjects will be recruited according to specific inclusion criteria after completion of medical and dental history questionnaires. Patients will sign a consent form after being advised about the nature of the study.

The selection of patients will be made according of the criteria approved by the 1999 international world workshop for a classification system of periodontal diseases and conditions using five clinical parameters and full mouth or panoramic radiographs for diagnosis.

Subjects will be allocated into four groups:

* Chronic Periodontitis group (ChP): comprise 20 patients aged > 45 years and have presence of ≥2 non-adjacent sites per quadrant that were not first molars or incisors, with probing depth (PD) ≥5 mm, which bleed on gentle probing. The demonstrated radiographic bone loss ≥30% of the root length, patient with poor oral hygiene, the amount of accumulated plaque commensurate with the amount of clinical attachment level (CAL)
* Resistant Control group (R): comprise 20 age-sex matched patients who are > 45 years exhibit no signs of periodontal disease as determined by the absence of the evidence of interproximal (CAL ≤ 1mm), PD > 3 mm at any site, whole-mouth bleeding scores <10% and have no clinical signs of gingival inflammation .
* Aggressive Periodontitis group (AgP): comprise 20 patients who are aged < 35 years and diagnosed with rapid attachment loss with periodontal pocket depth (PD) > 4 mm around at least three teeth other than the first molars and incisors. Rapid bone destruction (>50%bone loss at diseased sites). Weak relationship between dental plaque and the severity of gingival inflammation.
* Young Control group (YC): comprise 20 age- and sex matched patients who are < 35 years and exhibit no signs of periodontal disease.

Clinical measurements:

A standard periodontal probe will be used for recording periodontal indices at six sites per tooth. The examined clinical parameters include bleeding on probing (BOP), plaque index (PI), clinical attachment loss (CAL) and periodontal pocket depth (PPD) and gingival index (GI).

Collection of samples

Subjects will be asked to refrain from brushing within 1 hour of sampling. (GCF) samples will be obtained using standard paper strips (Periocol strips, Oraflow, NY, USA). 6 samples from each individual (mesiofacial, distopalatal) sites from each examined tooth (incisor, premolar and molar) in the maxilla (Chapple et al. 2002). Strips will be put in PBS Buffer solution for 30 minutes then extracted and stored under liquid nitrogen.

Venous blood samples will be collected from the antecubital fossa and stored in lithium heparin tubes and allowed to stand for 30 minutes before being centrifuged at 1000 ×g for 30 minutes, samples will be aliquoted into cryogenic vials and will be stored under liquid nitrogen.

Laboratory studies:

* TBARS assay (HPLC) will be used to assess the malondialdihyde levels as a marker of oxidative stress.
* Griess reagent to assess nitric oxide levels as a marker of nitrosative stress.

ELIGIBILITY:
Inclusion criteria:

* Patients of Syrian descent
* Systemically healthy
* Have at least 20 teeth

Exclusion criteria:

* Periodontal treatment during the last three months,
* History of major systemic diseases
* Consumption of anti oxidant supplements, antibiotics, anti inflammatory or any other drugs in the last three months
* Smoking
* Alcohol consumption
* Pregnant and lactating women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 80 subjects will be invited to participate in this study from the patients referred to the Department of Periodontology, Faculty of Dentistry, University of Damascus.
  The study has been pproved by our local Review Board. Subjects will be recruited according to specific inclusion criteria after completion of medical and dental history questionnaires. Patients will sign a consent form after being advised about the nature of the study.
  The selection of patients will be made according of the criteria approved by the 1999 international world workshop for a classification system of periodontal diseases and conditions (Armitage 1999) using five clinical parameters and full mouth or panoramic radiographs for diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Nitric oxide levels in serum and gingival cervicular fluid | Within 24 hours after the collection of the serum and gingival fluid
  Griess reagent to assess nitric oxide levels as a marker of nitrosative stress.
Malondialdihyide levels in serum and gingival cervicular fluid | Within 24 hours after the collection of the serum and gingival fluid
  TBARS assay (HPLC) will be used to assess the malondialdihyde levels as a marker of oxidative stress.

SECONDARY OUTCOMES:
Bleeding on Probing (BOP) | One time assessment once sample recruitment has completed. This outcome will be assessed within one week before treatment provision
  A standard periodontal probe will be used for recording periodontal indices at six sites per tooth. The examined clinical parameters include bleeding on probing (BOP)
Plaque Index (PI) | One time assessment once sample recruitment has completed. This outcome will be assessed within one week before treatment provision
  A standard periodontal probe will be used for recording periodontal indices at six sites per tooth.
Clinical Attachment Loss (CAL) | One time assessment once sample recruitment has completed. This outcome will be assessed within one week before treatment provision
  A standard periodontal probe will be used for recording periodontal indices at six sites per tooth.
Periodontal Pocket Depth (PPD) | One time assessment once sample recruitment has completed. This outcome will be assessed within one week before treatment provision
  A standard periodontal probe will be used for recording periodontal indices at six sites per tooth.
Gingival Index (GI). | One time assessment once sample recruitment has completed. This outcome will be assessed within one week before treatment provision
  A standard periodontal probe will be used for recording periodontal indices at six sites per tooth.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Alasadi, DDS, Principal Investigator — MSc student, Department of Periodontology, University of Damascus Dental School; Ali Abou Sulaiman, DDS MSc Phd, Study Director — Senior Lecturer in Periodontics, University of Damascus Dental School, Damascus; Francoise Qarabit, BSc MSc PhD, Study Director — Senior Lecturer in Chemistry, Department of Chemistry, Faculty of Sciences, University of Damascus, Baramkeh, Damascus, Syria
Locations (1):
- Department of Periodontics, University of Damascus Dental School, Damascus, Rif-dimashq Governorate, Syria

REFERENCES:
- [Background] Abou Sulaiman AE, Shehadeh RM. Assessment of total antioxidant capacity and the use of vitamin C in the treatment of non-smokers with chronic periodontitis. J Periodontol. 2010 Nov;81(11):1547-54. doi: 10.1902/jop.2010.100173. Epub 2010 Jun 22. PMID 20569170
- [Background] Armitage GC. Development of a classification system for periodontal diseases and conditions. Ann Periodontol. 1999 Dec;4(1):1-6. doi: 10.1902/annals.1999.4.1.1. PMID 10863370
- [Background] Chapple IL, Matthews JB. The role of reactive oxygen and antioxidant species in periodontal tissue destruction. Periodontol 2000. 2007;43:160-232. doi: 10.1111/j.1600-0757.2006.00178.x. No abstract available. PMID 17214840
- [Background] Halliwell B. Reactive oxygen species in living systems: source, biochemistry, and role in human disease. Am J Med. 1991 Sep 30;91(3C):14S-22S. doi: 10.1016/0002-9343(91)90279-7. PMID 1928205
- [Background] Kinane DF. Causation and pathogenesis of periodontal disease. Periodontol 2000. 2001;25:8-20. doi: 10.1034/j.1600-0757.2001.22250102.x. No abstract available. PMID 11155179
- [Background] Sies H. Oxidative stress: oxidants and antioxidants. Exp Physiol. 1997 Mar;82(2):291-5. doi: 10.1113/expphysiol.1997.sp004024. PMID 9129943
- [Background] Wactawski-Wende J. Periodontal diseases and osteoporosis: association and mechanisms. Ann Periodontol. 2001 Dec;6(1):197-208. doi: 10.1902/annals.2001.6.1.197. PMID 11887465